CLINICAL TRIAL: NCT05168540
Title: Frequency, Consequences, and Determinants of Suboptimal Care in the Initial Care Pathway of Child Physical Abuse: a Confidential Prospective Population-based Study in the French Western Region
Brief Title: Frequency, Consequences, and Determinants of Suboptimal Care in the Initial Care Pathway of Child Physical Abuse
Acronym: DIAPED
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0092
Record Dates: First submitted 2021-09-02; First posted 2021-12-23 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2024-08

CONDITIONS: Physical Abuse
Keywords: Child physical abuse; suboptimality; care pathway; population-based study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — Children will be included on the occasion of an admission to pediatric unit, the emergency room, the intensive care unit or a consultation in a specialized unit for children at risk of abuse. Their primary care pathway will be analyzed.

SUMMARY:
Physical abuse is a significant cause of morbidity and mortality in the general child population. There are no data specific to the French child care and protection systems, and very few studies have examined the optimality of protective measures following a diagnosis of child physical abuse. the investigators propose to conduct a confidential, prospective, population-based study, in order to assess the frequency of suboptimal care, to describe the typology of suboptimal care, to assess the immediate consequences of suboptimal care on the health of the child, and to identify the determinants of suboptimal care.

DETAILED DESCRIPTION:
Each year, 4 to 16% of minors are reported to be physically abused in high-incomes countries. Physical abuse is a significant cause of morbidity and mortality in the general child population. American and Canadian studies have shown that the diagnosis of child physical abuse is often delayed, putting children at risk of recurrence of abuse before diagnosis. There are no data specific to the French child care and protection systems, and very few studies have examined the optimality of protective measures following a diagnosis of child physical abuse. A better understanding of the typology of suboptimal care, its consequences and its determinants would allow to propose targeted action plans to optimize the care pathway and thus reduce the risk of recurrence and morbimortality. the investigators therefore propose to conduct a confidential, prospective, population-based study with an expert committee in the jurisdiction of the Court of Appeal of Rennes, in order to assess the frequency of suboptimal care, to describe the typology of suboptimal care, to assess the immediate consequences of suboptimal care on the health of the child, and to identify the determinants of suboptimal care. This study will allow a multidisciplinary work (medical, social, educational and legal) around child physical abuse in order to set up, in a second time, interventional trials to reduce these delays and to build the first French regional registry of child physical abuse.

ELIGIBILITY:
Inclusion Criteria:

* Children under the age of six who are suspected victims of physical abuse that led to an alert from authorities: traumatic skin or mucosal injury, (burn, bruise, hematoma, wound, conjunctival hemorrhages), intraocular hemorrhages, hemotympanum, traumatic looking intracranial injury, fracture, traumatic intra-abdominal or intra-thoracic injury to hollow or solid organs, non-accidental drug intoxication. For feasibility reasons, children will be included on the occasion of an admission to pediatric unit, the emergency room, the intensive care unit or a consultation in a specialized unit for children at risk of abuse. Their primary care pathway will be analyzed. Children who died in pre-hospital care in a context of strongly suspected maltreatment will also be included.

Non-inclusion Criteria:

* Emotional abuse, sexual abuse or neglect, without apparent physical harm.
* Children who have not been the subject of an administrative or judicial report by the hospital team taking care of the child.

Exclusion Criteria:

Child with a traumatic injury without suspicion of abuse.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under the age of six who are suspected victims of physical abuse that led to an alert from authorities.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Frequency in percentage of suboptimal care pathways | 2 years
  The optimality of the care will be evaluated by 2 independent experts and blinded to the final diagnosis (abuse confirmed or not) and to the child's health outcome

SECONDARY OUTCOMES:
- Main typologies of suboptimal care | 2 years
  the failures identified in the care pathway will be classified according to a grid and analyzed by experts. experts will classify the care pathway as optimal, suboptimal possible or suboptimal certain
Determinants of suboptimal care | 2 years
  The expertise will classify the children's care pathway as: optimal, suboptimal certain and suboptimal possible. The study of the determinants of suboptimal care will be carried out by comparing the characteristics of the children, their injuries and the actors involved in their care in each of the 3 groups
Potential consequences of suboptimal care in death | 12 months
  Analysis of the consequences of suboptimality in the care pathway will be done by comparing the number of dead patients with suboptimal care pathway, those surviving with sequelae and those surviving without sequelae at ICU discharge and at 12 months.
Potential consequences of suboptimal care in hospitalization | 2 years
  Analysis of the consequences of suboptimality in the care pathway will be done by comparing the number of patients hospitalized with suboptimal care pathway versus non-hospitalized patients, adjusting for the same variables as for survival
Potential consequences of suboptimal care on recurrency of child abuse | 1 years
  Analysis of the consequences of suboptimality in the care pathway will be done by comparing the number of patients with suboptimal care pathway with recurrences of child abuse or hospitalizations at one year to those without recurrences or hospitalizations at one year.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No